CLINICAL TRIAL: NCT03095781
Title: Phase Ib Trial of Pembrolizumab and XL888 in Patients With Advanced Gastrointestinal Malignancies
Brief Title: Pembrolizumab and XL888 in Patients With Advanced Gastrointestinal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Exelixis (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Olatunji Alese, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00087397; NCI-2016-01594 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship3321-16 (Other: Emory University/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2017-03-22; First posted 2017-03-30 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma; Recurrent Colorectal Carcinoma; Recurrent Pancreatic Carcinoma; Stage III Colorectal Cancer; Stage III Pancreatic Cancer; Stage IIIA Colorectal Cancer; Stage IIIB Colorectal Cancer; Stage IV Colorectal Cancer; Stage IV Pancreatic Cancer; Stage IVA Colorectal Cancer; Stage IVA Pancreatic Cancer; Stage IVB Colorectal Cancer; Stage IVB Pancreatic Cancer; Unresectable Pancreatic Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms | interventions — XL 888; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, XL888) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and XL888 PO on days 1, 4, 8, 11, 15, and 18. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: XL888; Biological: Pembrolizumab

INTERVENTIONS:
Drug: XL888 — Given PO
  Other Names: Heat Shock Protein 90 Inhibitor XL888; Hsp90 Inhibitor XL888
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase Ib trial studies the side effects and best dose of Hsp90 inhibitor XL888 when given together with pembrolizumab in treating patients with advanced gastrointestinal cancer that has spread to other places in the body. XL888 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as pembrolizumab, may block tumor growth in different ways by targeting certain cells. Giving XL888 with pembrolizumab may work better in treating patients with gastrointestinal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the recommended phase II dose for the combination of XL888 and pembrolizumab.

SECONDARY OBJECTIVES:

I. Define the toxicity profile of the combination of XL888 and pembrolizumab.

II. Evaluate the activity of the combination of XL888 and pembrolizumab in previously treated patients with gastrointestinal tumors.

TERTIARY OBJECTIVE:

I. Evaluate the effect of the combination on the immune profile in the serum and in tumor biopsies.

OUTLINE: This is a dose-escalation study of Hsp90 inhibitor XL888.

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and XL888 orally (PO) on day 1, 4, 8, 11, 15, and 18. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IV or locally advanced unresectable gastrointestinal adenocarcinomas (gastric, gastroesophageal junction [GEJ], cholangiocarcinoma, hepatocellular, pancreas, colorectal, small intestinal tumors) who have failed at least one prior therapy (dose escalation phase)
* Patients with pancreatic adenocarcinoma; patients must have histologic diagnosis and either locally advanced unresectable or metastatic disease that has failed at least one standard regimen; eight patients must have tumors that are accessible for biopsy and sign the informed consent for paired biopsy study (dose escalation phase, arm A)
* Patients with colorectal adenocarcinoma; patients must have histologic diagnosis and either locally advanced unresectable or metastatic disease and have previously received oxaliplatin, irinotecan, and fluoropyrimidine; eight patients must have tumors that are accessible for biopsy and sign the informed consent for paired biopsy study (dose escalation phase, arm B)
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) ≥ 1,500 cells/µL
* Platelets ≥ 100,000 cells/µL
* Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) ≥ 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x ULN OR ≤ 5 x ULN for subjects with liver metastases
* Albumin ≥ 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active tuberculosis (TB) (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or history of severe allergic or hypersensitivity reactions to excipients (e.g., polyethylene glycol [PEG] 300 and polysorbate 80)
* Clinically significant cardiovascular disease or peripheral vascular (e.g. myocardial infarction, unstable angina within 6 months of study entry), symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia requiring medications, baseline corrected QT (QTc) > 450 msec or previous history of QT prolongation while taking other medications
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has known substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-programmed death (PD)-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of the combination of XL888 and pembrolizumab as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Cycle length 21 days. Outcome determined on day 22 (after completion of cycle 1)
  Summary statistics will be presented. Toxicities will be presented as worst toxicity per patient and will be reported as percent toxicity.

SECONDARY OUTCOMES:
Overall response rate as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to 2 years after cycle 1, day 1. Cycle length is 21 days.
  RECIST version 1.1 will be used in this study for assessment of tumor response. While either CT or MRI may be utilized, as per RECIST 1.1, CT is the preferred imaging technique in this study.
Overall survival | Up to 1 year after cycle 1, day 1. Each cycle is 21 days.
  Once a subject experiences confirmed disease progression or starts a new anti-cancer therapy, the subject moves into the survival follow-up phase and should be contacted by telephone every 12 weeks to assess for survival status until death, withdrawal of consent, or the end of the study, whichever occurs first.
Progression free survival | Up to 6 months after cycle 1, day 1. Each cycle is 21 days
  Summary statistics will be presented.
Response duration as assessed by RECIST 1.1 | Up to 2 years after cycle 1, day 1. Each cycle is 21 days.
  Summary statistics will be presented.

OTHER OUTCOMES:
Immune profile effects of pembrolizumab and Hsp90 inhibitor XL888 assessed in serum and tumor biopsies | Up to 2 years after cycle 1, day 1. Each cycle is 21 days.
  Summary statistics will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Diab, MD, Principal Investigator — Emory University/Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

DOCUMENTS (1):
  • Informed Consent Form (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT03095781/ICF_000.pdf